CLINICAL TRIAL: NCT03539029
Title: Surgical Versus Conservative Treatment of Weber B1 Fracture: Functional Outcome Using Gait Analysis
Acronym: WEBER
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00513
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Ankle Fracture - Lateral Malleolus
MeSH Terms: conditions — Ankle Fractures | interventions — Surgical Procedures, Operative; Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: age and sex matched healthy control persons
- Surgery: patients with ankle fracture treated surgically
  Interventions: Procedure: Surgery
- Conservative treatment: patients with ankle fracture treated conservatively
  Interventions: Procedure: Conservative treatment

INTERVENTIONS:
Procedure: Surgery — Surgical fracture fixation
  Groups: Surgery
Procedure: Conservative treatment — immobilisation with plaster cast
  Groups: Conservative treatment

SUMMARY:
The decision whether to operate an ankle fracture or not is often highly dependent on the surgeon's individual judgment. There is consensus that non-displaced Weber A-type fractures rarely require operative treatment, and that Weber C-type or grossly displaced fractures are unstable and therefore require surgery. The decision for appropriate treatment is less clear for minimally displaced Weber B-type ankle fractures, and especially Weber B1 fractures are treated either surgically or conservatively at our clinic.

Conservative management of ankle fractures generally comprises immobilisation in a below-knee VacoPed or cast for six weeks to stabilise the fracture and allow osseous and soft tissue healing. Surgical treatment involves the reduction (if displaced) of the fractured fragments and fixation using various devices such as metal plates, screws, or intramedullary rods. While patients show changes in plantar pressure distribution during gait 18 months after surgical treatment of ankle fractures, to date the functional outcome regarding ankle joint mechanics during daily activities are unknown. Understanding gait function is important because compromised function may not only limit a persons daily activities but also may lead to secondary conditions such as osteoarthritis at the ankle or at adjacent joints.

The primary objective is:

• To compare differences in hindfoot and forefoot kinematics between level and uphill treadmill walking in relation to passive range of motion

The secondary objectives are:

* To compare ankle biomechanics during overground walking and level and uphill treadmill walking between patients with Weber B1 fracture treated either surgically or conservatively and healthy control persons.
* To determine the relationship between passive ankle range of motion, lower leg muscle strength and dynamic ankle range of motion.
* To determine the relationship between lower leg muscle strength and balance.
* To determine the relationship between dynamic range of motion and the Foot and Ankle Outcome Score.

DETAILED DESCRIPTION:
At the initial assessment, written informed consent will be obtained before participants will undergo a clinical exam (inspection and palpation of the foot, measurement of bilateral passive ankle range of motion). All participants will complete the Foot and Ankle Outcome score and the EQ-5D-5L health questionnaire to obtain pain and functional scores. Participants will be able to familiarize with treadmill walking at their preferred walking speed. Surface electrodes will be placed bilaterally over the tibialis anterior, gastrocnemius medialis and lateralis, soleus, and peroneus longus. Isokinetic muscle strength in ankle plantarflexion/ dorsiflexion will be tested using the Biodex system 4 Pro. Reflective surface markers will be placed bilaterally on anatomic landmarks according to the PlugIn Gait model9 and a specific foot model. These markers are seen by 8 Vicon cameras. Data for a standing reference trial will be collected, and participants will be asked to walk back and forth on a flat walkway until three valid left and right steps will be recorded (force plate hit centrally, approximately 10 minutes). Then, they will be asked to balance on one leg for 30 seconds per leg. Participants will be asked to stand on the treadmill (h/p cosmos, Zebris), and they will perform three single-limb heel rises with each leg while kinematic, electromyography (EMG), and pressure data will be measured. Participants will then walk barefoot for 2 minutes at 0% slope while kinematic, EMG, and pressure data will be recorded. Subsequently, the treadmill incline will be increased to 15%, and data for 2 minutes walking at this slope will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Surgical or conservative treatment after lateral malleolar fracture
* ≥12 months follow-up

Exclusion Criteria:

* Neuromuscular disorders affecting gait
* Additional pathologies that influence the mobility of the ankle joint
* Bilateral trauma at presentation
* Persistent use of walking aids
* Inability to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 20 patients with Weber B1 treated surgically; 20 patients with Weber B1 treated conservatively; 20 age and sex matched healthy control persons
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
3D hindfoot and forefoot range of motion during level and uphill walking | Baseline
  assessed in degrees as max plantarflexion to max dorsiflexion of the ankle using marker and camera based motion capture

SECONDARY OUTCOMES:
single leg balance | Baseline
  length of center of pressure during 30sec single leg stance measured in mm
ankle power | Baseline
  dynamic ankle power during walking measured in Nm/s
Isokinetic strength in plantarflexion, dorsiflexion, inversion, and eversion | Baseline
  Max moment assessed using a Biodex measured as Nm
Lower leg muscle activation | Baseline
  Max electromyographic signal intensity measured in mV
clinical outcome | Baseline
  assessed using the Foot and Ankle Outcome score (100 - no problems, 0 - extreme problems)
Health related quality of life | Baseline
  assessed using the EQ-5D-5L health questionnaire (100 - best healthy you can imagine; 0 - worst health you can imagine)
Pain in the ankle joint | Baseline
  assessed using a 15 cm visual analogue scale converted to 0 to 100 scale (0 - no pain; 100 - worst pain imaginable)
heel rise performance | Baseline
  To assess the single-limb heel rise ability, participants will complete three single-limb heel rise to maximum possible height. Heel rises will be performed with straight knees

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Mündermann, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided